CLINICAL TRIAL: NCT05388253
Title: Comparison of Static Stretching and Deep Kneading Massage Among Plantar Fasciitis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/508
Record Dates: First submitted 2022-05-05; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Stretching Among Plantar Fasciitis Patients (Experimental): Using Static Stretching exercises
  Interventions: Behavioral: Static Stretching
- Deep Kneading Massage Among Plantar Fasciitis Patients (Experimental): Using Deep Kneading Massage technique
  Interventions: Behavioral: Deep Kneading Massage

INTERVENTIONS:
Behavioral: Static Stretching — Using Static Stretching exercises
  Arms: Static Stretching Among Plantar Fasciitis Patients
Behavioral: Deep Kneading Massage — Using Deep Kneading Massage technique
  Arms: Deep Kneading Massage Among Plantar Fasciitis Patients

SUMMARY:
Comparison of Static Stretching and Deep Kneading Massage Among Plantar Fasciitis Patients

DETAILED DESCRIPTION:
To find out the better type of intevention in Static Stretching and Deep Kneading Massage for the betterment of Plantar Fasciitis Patients

ELIGIBILITY:
Inclusion Criteria:

* A person with phytoplitis by a doctor, physiotherapist or orthopedic surgeon.
* Determine the patient's age between 40 and 60 years.
* The patient's fracture, fracture, most cancers and various metabolism disorders are not used. Male and female victims can be involved.

Exclusion Criteria:

* Inflammatory arthritis patients.
* Nerve distortions
* Another disease caused in the case of March.
* Patients with various basic muscle problems and the effects of red science
* Does not use the patient's latest records and footprint.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Static Stretching Among Plantar Fasciitis Patients | 6 Months
  32 participants in Static stretches are those in which you stand, sit or lie still and hold a single position for a period of time, up to about 45 seconds with Visual Analogue Scale

SECONDARY OUTCOMES:
Deep Kneading Massage Among Plantar Fasciitis Patients | 6 Months
  32 participants in Deep-kneading massage is a technique which is used in relaxing relieving muscle strain and neck, back, shoulder, abdominal, leg and foot pain with Foot and Ankle Ability Measure (FAAM)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospitals, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No